CLINICAL TRIAL: NCT04042909
Title: Using Counter Attitudinal Advocacy to Change Drinking Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Houston (Other)
Responsible Party: Principal Investigator, Kate Carey, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1809002214; R01AA025043 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Drinking; Alcohol Abuse
Keywords: brief intervention; college students
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Counter Attitudinal Advocacy (Experimental): Participants in this arm will articulate ways to avoid alcohol-related consequences using self-generated protective strategies and publicly state those strategies.
  Interventions: Behavioral: Counter Attitudinal Advocacy
- Personalized Normative Feedback (Active Comparator): Participants in this arm will view personalized normative feedback regarding their 1) own drinking quantity and frequency of drinking, 2) perceptions of typical drinking by same-sex students' on campus (i.e., perceived descriptive norms), and 3) actual drinking rates by same-sex students' on campus (i.e., actual descriptive norms).
  Interventions: Behavioral: Personalized Normative Feedback
- Assessment-only Control (No Intervention): Participants in this arm will not receive any intervention.

INTERVENTIONS:
Behavioral: Counter Attitudinal Advocacy — same as Counter Attitudinal Advocacy arm
  Other Names: CAA
  Arms: Counter Attitudinal Advocacy
Behavioral: Personalized Normative Feedback — same as Personalized Normative Feedback arm
  Other Names: PNF
  Arms: Personalized Normative Feedback

SUMMARY:
High volume drinking by young adults has proven resistant to change, so new approaches are needed. We adapt a theory-based attitude change strategy for use in alcohol prevention. This research tests the impact of brief writing and advocacy activities on subsequent drinking and negative consequences.

DETAILED DESCRIPTION:
The persistence of risky drinking among young adults in college calls for continued efforts to prevent harms related to alcohol. Many prevention interventions rely on a primary mechanism of change: correcting exaggerated drinking norms. We propose to test a novel prevention strategy targeting another mechanism of change: creating attitude-behavior dissonance. To date, attitude change activities have not been harnessed as a behavior change strategy for alcohol abuse prevention, so this study adapts counter-attitudinal advocacy (CAA) to the alcohol prevention context. The goals of the proposed research are to demonstrate (a) the utility of CAA to change high volume drinking and related consequences, (b) that attitude change and attitude-behavior dissonance mediates the CAA manipulation effect, and (c) that CAA-induced risk reduction is not inferior to an established intervention based on Personalized Normative Feedback (PNF). A pair of studies will be implemented across two sites. First surveys to document peer behaviors and normative perceptions (N = 500 at each site) will be conducted, in order to deliver accurate, campus-specific PNF. The next study consists of a randomized controlled trial (RCT) with 2 experimental conditions (CAA and PNF) and a 3rd assessment only control condition to determine the impact of CAA on alcohol outcomes. For the RCT, a total of 600 heavy drinking students who have endorsed alcohol-related negative consequences will be recruited. Alcohol outcomes will be assessed at 1-, 3-, and 6-month follow-ups to test hypotheses that, relative to assessment only control, the CAA manipulation will decrease alcohol consumption and consequences. We will also test the hypothesis that CAA condition will be no less efficacious than (i.e., not inferior to) the PNF condition. The RCT also allows tests of hypotheses about effect moderators and mediators. This study will demonstrate the generalizability of CAA activities to the alcohol prevention context, as well as their generalizability across demographically different settings. Implications for the public health include establishing the efficacy of a new approach for reducing high volume drinking and related consequences among young adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26
* Male or female student at Brown University or University of Houston
* Past month heavy episodic drinking (for men, >5 drinks in one day, for women >4 drinks in one day)
* At least two self-reported negative consequences from drinking in the past month

Exclusion Criteria:

* status as a second semester Senior

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 591 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate B Carey, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the investigators to ensure that it meets reasonable demands of scientific integrity.
Supporting Information: Study Protocol, ICF
Time Frame: Within one year of study completion
Access Criteria: to be determined

REFERENCES:
- [Derived] Carey KB, DiBello AM, Hatch MR, Weinstein AP, Neighbors C. Efficacy of counter-attitudinal advocacy and personalized feedback for heavy-drinking college students. J Consult Clin Psychol. 2025 May;93(5):357-368. doi: 10.1037/ccp0000949. Epub 2025 Mar 13. PMID 40080603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Counter Attitudinal Advocacy | Personalized Normative Feedback | Assessment-only Control
Started | 194 | 197 | 200
Completed | 191 | 196 | 200
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — duplicate cases | 2 | 0 | 0
Not completed — technical problem | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counter Attitudinal Advocacy | Personalized Normative Feedback | Assessment-only Control | Total
Number analyzed (Participants) | 191 | 196 | 200 | 587
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (1.4) | 19.9 (1.7) | 20.0 (1.7) | 19.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 124 | 126 | 369
  Male | 72 | 72 | 74 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 43 | 47 | 136
  Not Hispanic or Latino | 145 | 153 | 153 | 451
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 3 | 7
  Asian | 46 | 47 | 44 | 137
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 20 | 13 | 49
  White | 80 | 95 | 93 | 268
  More than one race | 24 | 16 | 27 | 67
  Unknown or Not Reported | 22 | 17 | 20 | 59
Region of Enrollment [Number; unit: participants]
  United States | 191 | 196 | 200 | 587
Drinks per week [Mean (Standard Deviation); unit: drinks per week] — A sum of the number of standard drinks reported across the 7 days of a typical week in the last month.
  drinks per week | 9.9 (6.2) | 9.8 (5.9) | 10.0 (7.8) | 9.9 (6.7)
Alcohol problems [Mean (Standard Deviation); unit: problems] — Count of alcohol problems endorsed in the last month, using the 48-item Young Adult Alcohol Consequences Questionnaire; the total score ranges from 0-48 and higher scores indicate more problems experienced in the past 30 days.
  problems | 11.1 (7.0) | 12.0 (7.6) | 11.5 (7.2) | 11.5 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Week as Assessed by the Daily Drinking Questionnaire
Description: Number of standard drinks consumed in a typical week over the past 30 days; scores can range from zero but have no upper limit as they are counts of drinks
Time Frame: 6-month follow up
Population: Participants were included in this analysis if they provided drinks per week data at the 6-month follow-up
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Counter Attitudinal Advocacy | Personalized Normative Feedback | Assessment-only Control
Number analyzed (Participants) | 178 | 177 | 188
drinks per week | 6.8 (7.6) | 6.0 (5.2) | 7.1 (6.8)
Statistical Analysis 1: Comparison: Counter Attitudinal Advocacy vs Assessment-only Control; Our main hypothesis is that, relative to Assessment-Only control, the Counter Attitudinal Advocacy intervention will decrease alcohol consumption (drinks per week) from baseline to 6-months; Test type: Superiority; p = .646, Regression, Linear — This is the p-value of the CAA vs AO factor in the model; We used linear regression, controlling for baseline value of outcome and sex, to determine change in the outcome as a function of condition; beta coefficient = -0.309, 95% CI 2-sided [-1.632 to 1.013], Standard Error of Mean 0.690

2. Primary Outcome: Alcohol-related Consequences as Assessed by the Young Adult Alcohol Consequences Questionnaire
Description: The Young Adult Alcohol Consequences Questionnaire is a checklist of 48 different consequences that could be experienced over the past 30 days; the total score ranges from 0-48; higher scores indicate more problems experienced in the past 30 days
Time Frame: 6-month follow up
Population: Participants were included if they provided data at the 6 month follow-up
Measure: Mean (Standard Deviation); unit: problems
Arm/Group | Counter Attitudinal Advocacy | Personalized Normative Feedback | Assessment-only Control
Number analyzed (Participants) | 178 | 180 | 188
problems | 6.4 (7.0) | 7.2 (7.4) | 8.3 (8.6)
Statistical Analysis 1: Comparison: Counter Attitudinal Advocacy vs Assessment-only Control; Our main hypothesis is that, relative to Assessment-Only control, the Counter Attitudinal Advocacy intervention will decrease alcohol problems from baseline to 6-months; Test type: Superiority; p = .014, Regression, Linear; We used regression, controlling for baseline value of outcome and sex, to determine pre-post change in the outcome as a function of condition; beta coefficient = -1.90, 95% CI 2-sided [-3.41 to -0.39], Standard Error of Mean 0.77

ADVERSE EVENTS:
Time Frame: through study completion, an average of 12 months.
Arm/Group | Counter Attitudinal Advocacy | Personalized Normative Feedback | Assessment-only Control
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/196 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/196 | 0/200
Other Adverse Events (participants affected / at risk) | 0/191 | 0/196 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04042909/Prot_SAP_ICF_000.pdf